CLINICAL TRIAL: NCT02339870
Title: Caring for Caregivers: Increasing Cancer Caregiver Wellbeing and Comforting Sensitivity
Brief Title: Expressive Writing in Improving the Wellbeing or Comforting Capacity of Caregivers of Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9216; NCI-2014-02511 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9216 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-12-30; First posted 2015-01-16 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Caregiver
MeSH Terms: interventions — Psychiatric Rehabilitation; Caregivers

ARMS (3):
- Arm I (expressive disclosure) (Experimental): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about their emotions pertaining to managing and providing care for the cancer patient.
  Interventions: Other: Psychosocial Support for Caregiver; Other: Questionnaire Administration
- Arm II (benefit finding) (Experimental): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about any benefits that have arisen because of the cancer diagnosis.
  Interventions: Other: Psychosocial Support for Caregiver; Other: Questionnaire Administration
- Arm III (control) (Sham Comparator): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about an emotionally neutral topic.
  Interventions: Other: Questionnaire Administration; Other: Sham Intervention

INTERVENTIONS:
Other: Psychosocial Support for Caregiver — Complete expressive disclosure writing
  Arms: Arm I (expressive disclosure)
Other: Psychosocial Support for Caregiver — Complete benefit finding writing
  Arms: Arm II (benefit finding)
Other: Questionnaire Administration — Ancillary studies
Other: Sham Intervention — Complete writing on an emotionally neutral topic
  Arms: Arm III (control)

SUMMARY:
This randomized clinical trial studies expressive writing in improving the wellbeing or comforting capacity of caregivers of patients with cancer. Expressive writing is a type of intervention that asks people to write about important topics (in this case participants' experience with their spouses'/partners' cancer) and their emotions/feelings surrounding them. Expressive writing, including benefit finding and traumatic disclosure, may be a type of at-home-therapy that caregivers can utilize in an attempt to increase their own wellbeing, offer better comfort to cancer patients, and by association, help cancer patients cope with and manage the cancer experience.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether one, or both, types of expressive writing impact spouses of cancer survivors' reported emotional wellbeing and reported ability to provide comfort as compared to a control group.

OUTLINE: Patients are randomized to 1 of 2 arms or assigned to a control arm.

ARM I (EXPRESSIVE DISCLOSURE): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about their emotions pertaining to managing and providing care for the cancer patient.

ARM II (BENEFIT FINDING): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about any benefits that have arisen because of the cancer diagnosis.

ARM III (CONTROL): Participants complete an anonymous 20 minute writing exercise at home on their computer once per week for 2 weeks (days 2, 9, and 16 for a total of 3 sessions). Participants write about an emotionally neutral topic.

After completion of study, participants are followed up at day 17.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a spouse or domestic partner of a cancer survivor and will be recruited via the Hematopoietic Stem Cell Transplant Database at Fred Hutchinson Cancer Research Center (FHCRC)
* Participants must have been in their spousal relationship for at least the past 1 year

Exclusion Criteria:

* If participants are unable to access a computer they will be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in comforting sensitivity (i.e. quality of social support), measured through writing exercise and anonymous online survey | Baseline to day 17
  Will be reported pre- to post-test for both treatment groups compared to the control group. Repeated measures analysis of variance (ANOVA) within/between interaction will be used.
Change in comforting sensitivity (support quality), measured through writing exercise and anonymous online survey | Baseline to day 17
  Compared between women and men in both treatment groups using paired samples t-test.
Change in degree of stress pre- to post-test in predicting an increase in comforting strategies, measured through writing exercise and anonymous online survey | Up to day 17
  Will be analyzed using multiple linear regression.
Change in emotion regulation over time, measured through writing exercise and anonymous online survey | Baseline to day 17
  Will be compared between traumatic disclosure participants and the control group and between benefit finding participants and the control group using repeated measures ANOVA within/between interaction.
Change in stress, measured through writing exercise and anonymous online survey | Baseline to day 17
  Will be compared between women and men in both treatment groups using paired samples t-test.
Change in stress, perceived burden, and emotion regulation over time, measured through writing exercise and anonymous online survey | Baseline to day 17
  Will be compared between traumatic disclosure participants and the control group and between benefit finding participants and the control group using repeated measures ANOVA within/between group interaction.
Change in use of cognitive mechanism words in expressive writing in predicting significantly higher increases in comforting sensitivity (support quality), measured through writing exercise and anonymous online survey | Baseline to day 17
  Will be analyzed using multiple linear regression.
Changes in emotion regulation in predicting an increase in comforting strategies, measured through writing exercise and anonymous online survey | Up to day 17
  Will be analyzed using multiple linear regression.
Degree of stress, perceived burden, and emotion regulation in predicting comforting sensitivity (i.e. social support quality), measured through writing exercise and anonymous online survey | Up to day 17
  Analyzed using linear multiple regression.
Post-test emotion regulation scores, measured through writing exercise and anonymous online survey | Up to day 17
  Compared between traumatic disclosure and benefit finding groups using post-hoc analyses of repeated measures ANOVA.
Use of emotion-related words in predicting differences in comforting sensitivity (support quality), measured through writing exercise and anonymous online survey | Up to day 17
  Will be analyzed using multiple linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Harvey J, Berndt M. Cancer caregiver reports of post-traumatic growth following spousal hematopoietic stem cell transplant. Anxiety Stress Coping. 2021 Jul;34(4):397-410. doi: 10.1080/10615806.2020.1845432. Epub 2020 Nov 15. PMID 33190518
- [Derived] Harvey J, Sanders E, Ko L, Manusov V, Yi J. The Impact of Written Emotional Disclosure on Cancer Caregivers' Perceptions of Burden, Stress, and Depression: A Randomized Controlled Trial. Health Commun. 2018 Jul;33(7):824-832. doi: 10.1080/10410236.2017.1315677. Epub 2017 May 3. PMID 28467137